CLINICAL TRIAL: NCT06960278
Title: Effect of Alum Stone Containing Mucosal Adhesive Patches on Healing of Recurrent Aphthous Stomatitis: A Randomized Double-blinded Placebo-controlled Clinical Trial
Brief Title: Effect of Alum Stone Containing Mucosal Adhesive Patches on Healing of Recurrent Aphthous Stomatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Of Anbar (Other)
Responsible Party: Principal Investigator, Marwan Mahmood Saleh, Marwan Mahmood Saleh, University Of Anbar
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UAnbar
Record Dates: First submitted 2025-02-15; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Aphthous Stomatitis, Recurrent; Aphthous Stomatitis; Aphthous Ulcer
Keywords: Alum stone; aphthous ulcer; mucosal adhesive patches
MeSH Terms: conditions — Sutton disease 2; Stomatitis, Aphthous

STUDY DESIGN:
Intervention Model Description: In this study one hundred female, aged between twenty-two and thirty years, reported multiple oral aphthous ulcers. The evaluation of recurrent aphthous stomatitis (RAS) was performed by an oral medicine specialist, who relied on the clinical manifestations of the condition. The experimental group was administered 1x1cm mucosal patches containing alum stone at a concentration of 7%, whereas the control group was given placebo patches without any active medication. Size of aphthous lesions and degree of pain assessed at days 1, 3, and 5. Statistical analysis was performed with repeated measures ANOVA using R software
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A Randomized Double-blinded Placebo-controlled Clinical Trial (Placebo Comparator): The experimental group was administered 1x1cm mucosal patches containing alum stone at a concentration of 7%, whereas the control group was given placebo patches without any active medication
  Interventions: Procedure: Size of aphthous lesions and degree of pain assessed at days 1, 3, and 5.; Procedure: Control
- Control (Experimental)
  Interventions: Procedure: Size of aphthous lesions and degree of pain assessed at days 1, 3, and 5.; Procedure: Control
- Placebo (Placebo Comparator): hundred female from the patients of oral diagnosis clinic in college of dentistry and from the privet clinic
  Interventions: Device: ALUMSTONE

INTERVENTIONS:
Procedure: Size of aphthous lesions and degree of pain assessed at days 1, 3, and 5. — Size of aphthous lesions and degree of pain assessed at days 1, 3, and 5.
  Arms: A Randomized Double-blinded Placebo-controlled Clinical Trial; Control
Procedure: Control — The dimensions of the lesion were measured by oral medicine specialists using a flexible ruler
  Arms: A Randomized Double-blinded Placebo-controlled Clinical Trial; Control
Device: ALUMSTONE — alum administration via adhesive patches on the healing process of aphthous ulcers
  Arms: Placebo

SUMMARY:
The evaluation of recurrent aphthous stomatitis (RAS) was performed by an oral medicine specialist, who relied on the clinical manifestations of the condition. The experimental group was administered 1x1cm mucosal patches containing alum stone at a concentration of 7%, whereas the control group was given placebo patches without any active medication. Size of aphthous lesions and degree of pain assessed at days 1, 3, and 5. Statistical analysis was performed with repeated measures ANOVA using R software.

DETAILED DESCRIPTION:
The study's results indicated that the utilization of alum stone in mucosal adhesive patches yielded significant reductions in size of aphthous lesions and degree of pain.

ELIGIBILITY:
Inclusion Criteria: individuals who had a history of RAS, with oral ulceration occurring at least once a month and persistent oral ulceration being present in the majority of patients. Additionally, individuals with mild aphthous ulcer, characterized by ulcer development lasting fewer than three days, were also included.

-

Exclusion Criteria: Exclusion criteria encompassed the following: Pregnancy or lactation, systemic disorders linked to aphthous ulcers, such as Crohn's disease, Reiter's syndrome, and people who smoke or use cigarettes. Participants who were getting pharmacological therapy for fungal or viral infections, as well as those who were taking non-steroidal anti-inflammatory drugs, subjects with recent oral surgery, and those with fixed orthodontic appliances or retainers near the ulcer were not recruited for the study

-

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Lesion Size | 1, 3, 5 day

CONTACTS AND LOCATIONS:
Locations (1):
- Iraq, Anbar, Ramadi, 72300, Anbar, Al-Anbar Governorate, Iraq

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10808270/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24790718/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16120136/